CLINICAL TRIAL: NCT05460702
Title: Evaluation of the Relationship Between Stage I-II Breast Cancer Subtypes and Soluble Immune Checkpoints
Brief Title: Relationship Between Breast Cancer Subtypes and Immune Checkpoints
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ufuk Oguz Idiz, Assoc. Prof. MD. PhD, Istanbul Training and Research Hospital
Other Study IDs: Breast immune checkpoint
Record Dates: First submitted 2022-07-09; First posted 2022-07-15 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Immune Checkpoints
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Luminal A: Breast cancer patients with immunohistochemically luminal A
  Interventions: Diagnostic Test: Soluble immune checkpoints
- Luminal B: Breast cancer patients with immunohistochemically luminal B
  Interventions: Diagnostic Test: Soluble immune checkpoints
- Triple negative: Breast cancer patients with immunohistochemically triple negative
  Interventions: Diagnostic Test: Soluble immune checkpoints
- Control: The absence of any pathology in the breasts of healthy volunteers by mammography and/or ultrasound
  Interventions: Diagnostic Test: Soluble immune checkpoints

INTERVENTIONS:
Diagnostic Test: Soluble immune checkpoints — Blood collection from breast cancer patients with stage I-II

SUMMARY:
Breast cancer is the most common type of cancer in women and the second most common cause of death after lung cancer. The luminal group A, which has the highest prevalence among breast cancers; It includes Her2-negative tumors with low proliferative activity, low mitotic rate and histological grade. The prognosis of patients with luminal A tumors is very good and metastases are mostly limited to bones. Luminal-B tumors have a more aggressive course. The most important difference of this group is that tumors have a high proliferation rate. The breakpoint between luminal A and B is generally accepted as less than 14% of tumor cells showing nuclear Ki67 expression immunohistochemically. In addition, approximately 30% of Her2-positive tumors are immunohistochemically in the luminal B phenotype.

Up or down regulation of immune checkpoints is observed to protect breast cancer cells from the anti-tumor responses of the immune system. There are few studies in the literature evaluating soluble immune checkpoints in breast cancer, and these studies did not evaluate soluble immune checkpoints according to the histopathological subtyping of breast cancer.

The aim of this study is to determine the relationship between Luminal A, Luminal B and triple negative breast cancer and soluble immune control points, and to guide possible potential immunotherapy treatments.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer in women and the second most common cause of death after lung cancer. Its prevalence in epidemiological studies is 22-26%, and the risk of mortality due to breast cancer is around 18%. While the classification of malignant breast tumors has traditionally been based on histological appearance, but recently the subtypes have been defined according to their molecular features. The different behavior of tumors in the luminal group led to the need to divide this group into subtypes as luminal A and B. The luminal group A, which has the highest prevalence among breast cancers; It includes Her2-negative tumors with low proliferative activity, low mitotic rate and histological grade. The prognosis of patients with luminal A tumors is very good and metastases are mostly limited to bones. Luminal-B tumors have a more aggressive course. The most important difference of this group is that tumors have a high proliferation rate. The breakpoint between luminal A and B is generally accepted as less than 14% of tumor cells showing nuclear Ki67 expression immunohistochemically. In addition, approximately 30% of Her2-positive tumors are immunohistochemically in the luminal B phenotype.

It is known that the immune system has an important role in tumor development or tumor destruction. Recent studies have shown that tumor cells acquire escape mechanisms to escape host immunity in the tumor microenvironment.

Immune checkpoints are important molecules that are on the agenda especially after receiving the Nobel Prize in 2018 and in revealing the relationship between cancer and the immune system. Programmed Cell Death Protein-1 (PD-1) and its ligand, PD-L1, is an immune checkpoint that acts by inhibiting T cell receptor signaling and auxiliary stimuli. T cell immunoglobulin and mucin domain 3 (TIM-3) are mostly expressed on interferon-γ producing T cells, Tregs, dendritic cells, B cells, macrophages, natural killer cells (NK) and mast cells.

Studies have reported that immune checkpoints are elevated in many cancer types and have a poor prognosis. Immune checkpoints have naturally soluble forms of receptors and ligands, and although they are important components of immune regulation, their exact mechanism of action has not yet been determined. There are many studies on the effectiveness of immune checkpoints, especially in cancer patients.

Up or down regulation of immune checkpoints is observed to protect breast cancer cells from the anti-tumor responses of the immune system. Although many studies have been conducted on immune checkpoints in recent years, a limited number of immune checkpoints expressed on the cell surface have been evaluated in these studies. Measurement of soluble immune control points is easier than those expressed on the surface, and many markers can be evaluated at the same time. There are few studies in the literature evaluating soluble immune checkpoints in breast cancer, and these studies did not evaluate soluble immune checkpoints according to the histopathological subtyping of breast cancer.

In this study, patients with breast masses detected in Istanbul Training and Research Hospital and Memorial Hizmet Hospital Breast Diseases outpatient clinic between April 2022 and September 2022 will constitute the population of the patient group. Volunteers who applied to the breast diseases outpatient clinic and who did not have any breast problems in their examinations will be included as the control group. The trucut biopsy pathology reports of the breast masses of the patients included in the study will be examined, and if breast cancer is detected, the clinical stage will be evaluated. Breast cancer patient with stage I-II will be divided into three groups immunohistochemically like as Luminal A, Luminal B and Triple negative.

After the diagnosis of breast cancer from the patients and the absence of any pathology in the breasts of healthy volunteers by mammography and/or ultrasound, 10 cc of blood will be drawn into the biochemistry tube, their serum will be separated by centrifugation and stored in a -80oC refrigerator. After the collection of all samples, the flow cytometric analysis will be performed and serum immune checkpoints will be measured.

The aim of this study is to determine the relationship between Luminal A, Luminal B and triple negative breast cancer and soluble immune checkpoints, and to guide possible potential immunotherapy treatments.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years,
* Patients with clinically and histopathologically proven Stage I-II breast cancer

Exclusion Criteria:

* Known immunodeficiency
* Having a primary malignancy other than breast cancer,
* Pregnancy,
* Patients younger than 18 years and older than 90 years,
* Patients who refused to participate in the study

Ages: 18 Years to 90 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Breast cancer patient with stage I-II
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Immune checkpoints | 2 weeks
  sCD25 (pg/ml), 4-1BB (pg/ml), B7.2 (pg/ml), Free Active TGF-β1 (pg/ml), CTLA-4 (pg/ml), PD-L1 (pg/ml), PD-1 (pg/ml), Tim-3 (pg/ml), LAG-3 (pg/ml), Galectin-9 (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Ufuk Oguz Idiz, Assoc.Prof., Principal Investigator — Istanbul Training and Research Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Training and Research Hospital, Istanbul
  - Memorial Hizmet Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gu D, Ao X, Yang Y, Chen Z, Xu X. Soluble immune checkpoints in cancer: production, function and biological significance. J Immunother Cancer. 2018 Nov 27;6(1):132. doi: 10.1186/s40425-018-0449-0. PMID 30482248
- [Result] Fang J, Chen F, Liu D, Gu F, Chen Z, Wang Y. Prognostic value of immune checkpoint molecules in breast cancer. Biosci Rep. 2020 Jul 31;40(7):BSR20201054. doi: 10.1042/BSR20201054. PMID 32602545
- [Result] Asano Y, Kashiwagi S, Takada K, Ishihara S, Goto W, Morisaki T, Shibutani M, Tanaka H, Hirakawa K, Ohira M. Clinical Significance of Expression of Immunoadjuvant Molecules (LAG-3, TIM-3, OX-40) in Neoadjuvant Chemotherapy for Breast Cancer. Anticancer Res. 2022 Jan;42(1):125-136. doi: 10.21873/anticanres.15466. PMID 34969718